CLINICAL TRIAL: NCT03297840
Title: Change in Mindfulness in Borderline Personality Disorder After Dialectic-behavioural Therapy (DBT): A Pre-post-comparison
Brief Title: Change in Mindfulness in Borderline Personality Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Katharina Bachmann (Other)
Responsible Party: Sponsor-Investigator, Katharina Bachmann, Psychologist Msc., University of Oldenburg
Organization: University of Oldenburg (Other)
Other Study IDs: Mindfullness in BPD
Record Dates: First submitted 2017-05-09; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Mindfulness; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment: Patients with Borderline Personality Disorder receiving DBT treatment. Measurement takes place at the beginning of the treatment and a second time after 12-weeks treatment.
  Interventions: Behavioral: Dialectical Behavioural Therapy (DBT)
- Waitlist: Patients with Borderline Personality Disorder on the waitlist for inpatient DBT treatment. Measurement takes place twice at baseline and after 12-weeks waiting.

INTERVENTIONS:
Behavioral: Dialectical Behavioural Therapy (DBT) — Inpatient Dialectical Behavioural Therapy (DBT) according to Linehan.
  Groups: Treatment

SUMMARY:
The current study aims to investigate the effect of dialectical behavioral therapy on mindfulness in patients with Borderline Personality Disorder. A treatment group will be compared to a waitlist control group.

DETAILED DESCRIPTION:
Participants will be recruited from the Dialectical-Behavioral-Therapy (DBT) unit. DBT is a treatment approach that has been shown to be effective in the treatment of Borderline Personality Disorder. DBT integrates different psychotherapeutic interventions as well as Mindfulness Meditation exercises. Mindfulness is a meditation practice that can improve present moment awareness. When applied as therapeutic intervention mindfulness meditation can help patients to stay with their attention in the present moment, to be aware what is happening in the here and now, and to better identify and regulate upcoming emotions.

The current observational study investigates changes in symptom severity and mindfulness skills during DBT treatment. A treatment group will be compared to a waitlist control group. The two groups are predefined by routine medical care.

Symptom severity and mindfulness skills will be assessed at baseline (before treatment or when accepted for the waitlist) and after 12-weeks. A within and between group analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Borderline Personality Disorder
* On the waitlist for DBT treatment or actually treated with DBT
* Not previously treated with DBT.

Exclusion Criteria:

* Severe psychiatric comorbidity e.g. psychosis, severe depression, suicidality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male and female BPD Patients from 18 to 60 years.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in mindfulness | Baseline and after 12-weeks
  Degree of mindfulness will be assessed by the Kentucky Inventory of Mindfulness Skills, German Version (KIMS-D). A within and between group comparison will be performed (treatment vs. waitlist).
Change in borderline symptom severity | Baseline and after 12-weeks
  Change in Borderline symptom severity is measured by the Borderline Symptom List (BSL 23). A within and between group comparison will be performed (treatment vs. waitlist).
Change in overall psychiatric symptom severity | Baseline and after 12-weeks
  Change in overall symptom severity is measured by the Change in symptomseverity is measured by the Symptom-Checklist-90®-Standard (SCL-90). A within and between group comparison will be performed (treatment vs. waitlist).
Change in severity in symptoms of depression | Baseline and after 12-weeks
  Change in overall symptom severity is measured by the Beck depression inventory (BDI). A within and between group comparison will be performed (treatment vs. waitlist).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Philipsen, Prof., Principal Investigator — Department of Psychiatry and Psychotherapy - University Hospital, University of Oldenburg, Oldenburg, Germany
Locations (1):
- Department of Psychiatry and Psychotherapy - University Hospital, University of Oldenburg, Bad Zwischenahn, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793